CLINICAL TRIAL: NCT02437656
Title: Phase II Study Evaluating the Efficacy of the Combination of Metformin to Neoadjuvant Radiochemotherapy in the Treatment of Locally Advanced Rectal Cancer.
Brief Title: Combination of Metformin to Neoadjuvant Radiochemotherapy in the Treatment of Locally Advanced Rectal Cancer (METCAP).
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Oscar Lambret (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: METCAP-1404; 2014-003687-20 (EudraCT Number)
Record Dates: First submitted 2015-05-05; First posted 2015-05-07 (Estimated); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Rectal Cancer
Keywords: Radiochemotherapy; Metformin; Rectal cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Metformin treatment (Experimental): J1 : dosimetric scan
  J3 : initiation of the Metformin therapy (at a dosage of 1700 mg / day)
  J10 : increasing the dose of Metformin (2550 mg / day) + initiation of the radiochemotherapy
  J44 : end of the radiochemotherapy
  Between J86 and J100 : surgery (discontinuation of the Metformin therapy 48 hours before surgery)
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — J3 - J10 (7 days minimum) : 850 mg 2 times / day
  J10 - 48h before surgery : 850 mg 3 times / day
  Other Names: Glucophage; Diabamyl; Stagid

SUMMARY:
Metformin is an oral antidiabetic of the biguanide class derived from galega officinalis. Historical cohort of patients with diabetes have shown that diabetics on Metformin had a better chance of survival than diabetics not on Metformin. These observations have led to in vitro studies of metformin on cancer cells. It was thus demonstrated that Metformin has anti-proliferative properties.

The aim of our study is to evaluate the efficacy of metformin in combination with neoadjuvant radiochemotherapy in the treatment of locally advanced rectal cancer.

DETAILED DESCRIPTION:
Patients eligible for the trial and having signed their consent to participate will undergo a dosimetric scan at baseline. 48 hours later (minimum), a Metformin therapy will be started at a dosage of 850 mg 2 times / day ( = 1700 mg / day). Seven days later (minimum) and up to 48 hours before surgery, the dosage of Metformin will be increased to 850 mg 3 times / day ( = 2550 mg / day). This very same day (J10), patients will start a radiochemotherapy. For 5 weeks, 5 days out of 7, patients will receive 800 mg/m² of Capecitabine 2 times / day (on morning and evening) ( = 1600 mg / m² / day) and a 3D irradiation or an Intensity-Modulated Radiation Therapy (IMRT) of a total dose of 50 Gy (5 sessions of 2 Gy per week). 6 to 8 weeks after completion of the chemoradiotherapy, surgery will be scheduled. It will consist of a tumor resection with total resection of the meso rectum.

Prior to the start of treatment, patients will have a clinical and a paraclinical examination and will undergo a laboratory examination. Once a week during the radiochemotherapy, patients will have a clinical examination and will undergo a laboratory examination. Three weeks after the end of the radiochemotherapy, patients will have a clinical examination. Before surgery, patients will have a clinical and a paraclinical examination. Finally, at the end of the study, patients will have a clinical examination.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with an adenocarcinoma of the low or middle rectum.
2. T3 or T4 stage (T evaluated by MRI and / or echo-endoscopy).
3. Absence of distant metastasis.
4. Patient requiring a radiochemotherapy.
5. Correct hematological conditions : Neutrophils ≥ 1500 G / L, platelets ≥ 100 000 G / L.
6. Age ≥ 18 years
7. Performance status (WHO) ≤ 2
8. Lactatemia ≤ Higher standard of the sampling laboratory.
9. For women of childbearing age, a contraceptive method is mandatory for the entire duration of the study.

Exclusion Criteria:

1. Other histologies such as squamous cell carcinoma, neuroendocrine tumors, melanomas, etc.
2. History of lactic acidosis.
3. Any diabetes (According to the WHO definition : fasting plasma glucose (FPG) > 1.26 g / L-1).
4. Ongoing antidiabetic treatment such as

   * Biguanides, hypoglycemic sulfamides, glinides, GLP-1 analogue, gliptins, alpha-glucosidase inhibitors
   * Insulin or insulin analogues
5. Hypersensitivity to capecitabine or to any of the excipients or to fluorouracil.
6. History of severe and unexpected reactions to a fluoropyrimidine therapy.
7. Patient with known deficiency to the dihydropyrimidine dehydrogenase (DPD).
8. Hypersensitivity to metformin or to any of the excipients.
9. Renal failure or impaired renal function (creatinine clearance < 60 ml / min).
10. Severe infection.
11. Acute or chronic disease which may cause tissue hypoxia such as heart or respiratory failure or recent myocardial infarction (< 6 months).
12. Hepatic insufficiency, acute alcohol intoxication, alcoholism.
13. Psychiatric inability to give consent.
14. Contraindication to radiation therapy and/or chemotherapy.
15. Treatment with sorivudine or its chemically related analogues, such as brivudine.
16. Patient under tutorship or guardianship.
17. Pregnant or breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-05; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
The efficacy will be assessed on the operative specimen by the complete histological response rate (absence of tumor cells : pCR). | within 30 days after surgery

SECONDARY OUTCOMES:
Toxicity will be assessed according to NCI-CTCAE v4.0. Grades ≥ 3 related to metformin will be collected by the clinician. | up to 30 days after the end of the treatments (metformin and radiochemotherapy)
Sphincter preservation rate and downstaging rate | within 30 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Xavier MIRABEL, MD, Principal Investigator — Centre Oscar Lambret
Locations (11):
- France (11):
  - Centre Marie Curie, Arras
  - Centre Pierre Curie, Beuvry
  - Centre Léonard de Vinci - SARL du pont Saint Vaast, Douai
  - Institut André Dutreix, Dunkirk
  - Centre Hospitalier, Lens
  - Clinique du Bois - Centre Bourgogne, Lille
  - Centre Oscar Lambret, Lille
  - Centre Galilée - Hôpital Privé La Louvière, Lille
  - Centre Gray, Maubeuge
  - Centre Joliot-Curie, Saint-Martin-Boulogne
  - Clinique des Dentellières, Valenciennes

IPD SHARING:
Plan to Share IPD: No